CLINICAL TRIAL: NCT04351360
Title: Pilot Study on Subjective Efficiency of Caffeine in ADCY5-related Dyskinesia
Brief Title: Pilot Study on Caffeine Efficiency in ADCY5-related Dyskinesia
Acronym: CAF-ADCY5
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C19-26; 2020-A00166-33 (Registry Identifier: 2020-A00166-33)
Record Dates: First submitted 2020-04-13; First posted 2020-04-17 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-04

CONDITIONS: Dyskinesias
Keywords: ADCY5 mutation
MeSH Terms: conditions — Dyskinesias

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Heterozygous mutations in the ADCY5 gene cause involuntary early-onset hyperkinetic movements. In addition, patients may have associated psychiatric disorders.There is currently no treatment. As the pathophysiology is linked to ADCY5 hyperactivity, the investigative team has treated patients with caffeine, an antagonist. The investigator wishes to interview patients on the effect of caffeine on their motor symptoms and their overall clinical condition, and on the possible existence of psychiatric comorbidities using phone questionnaires.

DETAILED DESCRIPTION:
Heterozygous mutations in the ADCY5 gene cause involuntary early-onset hyperkinetic movements. The phenotype combines chorea, dystonia and / or myoclonus with frequent facial involvement, axial hypotonia, fluctuations and / or episodes of paroxysmal dyskinesia which can be nocturnal and / or painful.

Many treatments have been tried, with no obvious efficacy. Two patients from the same family (a father and daughter) told investigators that caffeine had a dramatic effect on their paroxysmal episodes. They said that taking coffee would prevent episodes and reduce their duration (efficacy estimated at 80%), an effect specific to caffeine since it was reproduced by the ingestion of caffeine citrate capsules. Very interestingly, there is a rationale underlying this phenomenon. Indeed, caffeine is an antagonist of the adenosine A2A receptors (A2AR), receptors which activate ADCY5 and which are localized preferentially in striatal neurons expressing dopamine D2 receptors. As caffeine is an A2AR antagonist, it likely inhibits ADCY5, and therefore induces clinical improvement in patients with hyperactivity of this protein.

In addition, the investigative team noted anxiety in some of its patients, and the question of the presence of psychiatric disorders in ADCY5 patients was recently raised in the literature.

The investigative team wishes to collect standardized preliminary data by questioning patients on the effect of caffeine on their motor symptoms and their overall clinical state, and on the possible existence of psychiatric comorbidities using structured questionnaires which will be carried out by phone.

ELIGIBILITY:
Inclusion Criteria:

* Proven genetic diagnosis of ADCY5-related dyskinesia
* Caffeine intake
* Non opposition by the patient or the legal representatives if the patient is a minor.

No Exclusion Criteria.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ADCY5-related dyskinesia being actively treated, or who have been previously treated, with caffeine.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
Percentage of responders to caffeine | one hour
  the response being defined as an improvement of overall involuntary movements of 40% or more.

SECONDARY OUTCOMES:
Global change of involuntary movements ranging from 0 (no change) to 10 (disappearance of involuntary movements) | one hour
  evaluated by patients
Global clinical change ranging from 0 (no change) to 10 (normalization of the global clinical state) | one hour
  evaluated by patients
Change of the duration of paroxysmal episodes of movement disorders with caffeine | one hour
  evaluated by patients
Frequency change of paroxysmal episodes of movement disorders with caffeine | one hour
  evaluated by patients
Presence or absence of psychiatric symptoms | one hour
  according to the MINI (Mini International Neuropsychiatric Interview)

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie Meneret, Principal Investigator — APHP
Locations (1):
- Département de Neurologie Groupe Hospitalier Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen DH, Meneret A, Friedman JR, Korvatska O, Gad A, Bonkowski ES, Stessman HA, Doummar D, Mignot C, Anheim M, Bernes S, Davis MY, Damon-Perriere N, Degos B, Grabli D, Gras D, Hisama FM, Mackenzie KM, Swanson PD, Tranchant C, Vidailhet M, Winesett S, Trouillard O, Amendola LM, Dorschner MO, Weiss M, Eichler EE, Torkamani A, Roze E, Bird TD, Raskind WH. ADCY5-related dyskinesia: Broader spectrum and genotype-phenotype correlations. Neurology. 2015 Dec 8;85(23):2026-35. doi: 10.1212/WNL.0000000000002058. Epub 2015 Nov 4. PMID 26537056
- [Background] Friedman JR, Meneret A, Chen DH, Trouillard O, Vidailhet M, Raskind WH, Roze E. ADCY5 mutation carriers display pleiotropic paroxysmal day and nighttime dyskinesias. Mov Disord. 2016 Jan;31(1):147-8. doi: 10.1002/mds.26494. Epub 2015 Dec 21. No abstract available. PMID 26686870
- [Background] Lee KW, Hong JH, Choi IY, Che Y, Lee JK, Yang SD, Song CW, Kang HS, Lee JH, Noh JS, Shin HS, Han PL. Impaired D2 dopamine receptor function in mice lacking type 5 adenylyl cyclase. J Neurosci. 2002 Sep 15;22(18):7931-40. doi: 10.1523/JNEUROSCI.22-18-07931.2002. PMID 12223546
- [Background] Meneret A, Gras D, McGovern E, Roze E. Caffeine and the Dyskinesia Related to Mutations in the ADCY5 Gene. Ann Intern Med. 2019 Sep 17;171(6):439. doi: 10.7326/L19-0038. Epub 2019 Jun 11. No abstract available. PMID 31181574
- [Background] Vijiaratnam N, Newby R, Kempster PA. Depression and psychosis in ADCY5-related dyskinesia-part of the phenotypic spectrum? J Clin Neurosci. 2018 Nov;57:167-168. doi: 10.1016/j.jocn.2018.08.049. Epub 2018 Aug 30. PMID 30172639
- [Background] Yamada K, Kobayashi M, Kanda T. Involvement of adenosine A2A receptors in depression and anxiety. Int Rev Neurobiol. 2014;119:373-93. doi: 10.1016/B978-0-12-801022-8.00015-5. PMID 25175973
- [Result] Meneret A, Mohammad SS, Cif L, Doummar D, DeGusmao C, Anheim M, Barth M, Damier P, Demonceau N, Friedman J, Gallea C, Gras D, Gurgel-Giannetti J, Innes EA, Necpal J, Riant F, Sagnes S, Sarret C, Seliverstov Y, Paramanandam V, Shetty K, Tranchant C, Doulazmi M, Vidailhet M, Pringsheim T, Roze E. Efficacy of Caffeine in ADCY5-Related Dyskinesia: A Retrospective Study. Mov Disord. 2022 Jun;37(6):1294-1298. doi: 10.1002/mds.29006. Epub 2022 Apr 5. PMID 35384065